CLINICAL TRIAL: NCT02166580
Title: Comparison of the Non-invasive CNAP Pulse Pressure Variation With the Invasive Gold Standard
Brief Title: Accuracy of CNAP PPV Under General Anaesthesia
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, PD Dr. med. Jochen Renner, University Hospital Schleswig-Holstein
Other Study IDs: CNAP 2012_2
Record Dates: First submitted 2012-12-04; First posted 2014-06-18 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: General Anaesthesia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Noninvasive pulse pressure variation for the guidance of perioperative fluid therapy is compared with the gold standard of invasive measurements. Cardiac output is derived by the PICCO monitor.

Hypothesis: Noninvasive CNAP PPV predicts fluid responsiveness. A grey zone for the prediction of fluid responsiveness will be defined.

DETAILED DESCRIPTION:
Accuracy of PPV measured by two devices,PICCO and CNAP, is compared with the manually calculated PPV from the arterial line waveform. Established tests like passive leg raising and end-expiratory occlusion are used for prediction of fluid responsiveness. Intraoperative events like volume challenge are monitored.

ELIGIBILITY:
Inclusion Criteria:

* major surgery
* need for invasive arterial measurements

Exclusion Criteria:

* age under 18
* cardiac dysrhythmia
* vascular pathology at punction site

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major surgery with the need for invasive arterial pressure monitoring
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Cardiac output | 1, 2, 5, 10, 15 and 20 minutes after volume challange and
  Improvement of cardiac output dependent on PPV before volume challenge

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Renner, PD Dr., Principal Investigator — University Hospital Schleswig-Holstein, Departement of Anaesthesia and Intensive Care Medicine; Robert Hanss, Prof. Dr., Principal Investigator — University Hospital Schleswig-Holstein, Departement of Anaesthesia and Intensive Care Medicine
Locations (1):
- University Hospital, Schleswig-Holstein. Departement of Anaesthesiology and Intensive Care Medicine, Kiel, Germany

REFERENCES:
- [Derived] Renner J, Gruenewald M, Hill M, Mangelsdorff L, Aselmann H, Ilies C, Steinfath M, Broch O. Non-invasive assessment of fluid responsiveness using CNAP technology is interchangeable with invasive arterial measurements during major open abdominal surgery. Br J Anaesth. 2017 Jan;118(1):58-67. doi: 10.1093/bja/aew399. PMID 28039242